CLINICAL TRIAL: NCT06824116
Title: The Effect of Endurance Training on Exercise Tolerance, Motor Abilities, Cognitive Functions and Concentration of Selected Blood Biomarkers in Post-stroke Patients
Brief Title: The Effect of Endurance Training on Motor and Cognitive Functions and Concentration of Biomarkers in Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 378/21
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Ischemic; Stroke Patients
Keywords: stroke; cognitive functions; neurotrophins; neurological rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise low intensity (Active Comparator)
  Interventions: Behavioral: Exercise
- exercise moderate intensity (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Training on a bicycle ergometer was performed four times a week for 3 weeks for 45 min. The exercise intensity corresponded to 50%-60% of maximal oxygen uptake (VO2max).
  Arms: exercise low intensity
Behavioral: Exercise — Training on a bicycle ergometer was performed four times a week for 3 weeks for 45 min. The exercise intensity corresponded to 70 - 80% of maximal oxygen uptake (VO2max).
  Arms: exercise moderate intensity

SUMMARY:
The aim of this randomised experimental study is to test the effect of different intensities of aerobic exercise on neurotrophin concentration and functional and cognitive functions in post-stroke patients undertaking a single bout and 3-week exercise programme. The main questions to answer are:

1. What is effect of different intensities of aerobic exercise on functional abilities in post-stroke patients undertaking a 3-week aerobic exercise programme?
2. What is effect of different intensities of aerobic exercise on cognitive functions in post-stroke patients undertaking a 3-week aerobic exercise programme?
3. What is effect of different intensities of aerobic exercise on neurotrophin concentration in post-stroke patients undertaking a 3-week aerobic exercise programme?
4. What is effect of different intensities of 45-min single bout aerobic exercise on neurotrophin concentration in post-stroke patients?

The participants were randomly assigned to one of two groups: moderate-intensity continuous training on a bicycle ergometer and standard neurorehabilitation or low-intensity continuous training on a bicycle ergometer and standard neurorehabilitation. Training on a bicycle ergometer was performed four times a week for 45 min for 3 weeks. Each participant attended individual neurorehabilitation sessions 11 times per week (2 physical therapy sessions from Monday to Friday for 45 min each and 1 session on Saturday for 45 min) during the 3-week intervention.

Participants will have pre-tests and post-tests:

* blood samples collection (to measure level of brain-derived neurotrophic factor, glial cell derived neurotrophic factor, insulin-like growth factor, vascular-endothelial growth factor, irisin),
* body mass index
* The Graded Cycling Test with Talk Test
* 6-Minute Walk Test
* Rivermead Motor Assessment
* Barthel Index
* Addenbrooke's Cognitive Examination
* Vo2max
* Beck Depression Inventory

Researchers will compare two groups - moderate intensity continuous group and low intensity continuous group to see if there is a modulating effect of different intensities of exercise in participants' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 21-75 years,
* first episode of ischemic stroke confirmed by magnetic resonance imaging (MRI) or computed tomography (CT),
* able to walk for 4 m at a self-selected speed independently or with an assistive device (as needed),
* be in a stable clinical condition,
* able to communicate with investigators,
* provided written informed consent to participate in the study.

Exclusion Criteria:

* aphasia,
* an unstable cardiac status (e.g., evidence of significant arrhythmia or myocardial ischaemia),
* lower extremity claudication,
* weight-bearing pain >4/10,
* lower extremity spasticity (i.e., an Ashworth Scale score >2), other neurological conditions in addition to stroke,
* chronic degenerative or inflammatory diagnoses, malignancies, and visuospatial neglect.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Brain-derived neurotrophic factor | Before and after 3-week intervention; pre and post single bout of exercise in the first day of intervention
  Level of brain-derived neurotrophic factor in ng/ml
Glial cell derived neurotrophic factor | Before and after 3-week intervention; pre and post single bout of exercise in the first day of intervention
  Level of glial cell derived neurotrophic factor in ng/ml
Insulin-like growth factor | Before and after 3-week intervention; pre and post single bout of exercise in the first day of intervention
  Level of insulin-like growth factor in ng/ml
irisin | Before and after 3-week intervention; pre and post single bout of exercise in the first day of intervention
  Level of irisin in ng/ml
Vascular-endothelial growth factor A | Before and after 3-week intervention; pre and post single bout of exercise in the first day of intervention
  Level of Vascular-endothelial growth factor A in ng/ml
The Graded Cycling Test with Talk Test | Before and after 3-week intervention
  Cardiorespiratory fitness assessment with the Graded Cycling Test with Talk Test assess submaximal exercise in Watt. Higher Watt means better outcome.
Vo2max | Before and after 3-week intervention
  Physical performance assessment with Vo2max in mL/min/kg.
Six Minute Walk Test | Before and after 3-week intervention
  The 6 minute walking test assesses functional capacity during continuous walking on a 12-m ward hallway for 6 min. The test measures the distance a patient walks in 6 min.
Rivermead Motor Assessment | Before and after 3-week intervention
  Functional mobility among post-stroke patients was assessed with the Rivermead Motor Assessment, a performance-based measure in points. This later includes 38 items that cover three sections: gross function, leg and trunk and arm function. The total score ranges from 0 to 38 points. Higher scores indicate a higher degree of functional mobility.
Barthel Index | Before and after 3-week intervention
  The Barthel Index is a scale that measures an individual's functional outcomes. It consists of 10 items that assess activities of daily living, functional mobility, and gait. The score ranges from 0 to 100 points. The higher the score, the greater the individual's ability to self-care
Addenbrooke's Cognitive Examination | Before and after 3-week intervention
  Cognitive functions assessment with Addenbrooke's Cognitive Examination in points. Higher scores means better outcome.
Beck Depression Inventory | Before and after 3-week intervention
  Depressive symptoms assessment with Beck Depression Inventory in points. Higher scores means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiology, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No